CLINICAL TRIAL: NCT05195996
Title: Beta Blocker Effects on Patients With Traumatic Brain Injury
Brief Title: Beta Blocker Effects in Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2/2021ANESTH-4
Record Dates: First submitted 2021-12-02; First posted 2022-01-19 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Trauma, Brain
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propranolol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- beta blocker (Active Comparator): Will be given Propranolol 1mg in 10 ml distilled water intravenous every 6 hours for 48 hours
  Interventions: Drug: Propranolol
- placebo (Placebo Comparator): Will be given normal saline 10 ml every 6 hours for 48 hours
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Propranolol — intravenous propranolol for case patients
  Arms: beta blocker
Drug: Saline — intravenous saline for placebo
  Arms: placebo

SUMMARY:
The study will be conducted on polytrauma patient who are admitted from emergency room or postoperative with head trauma to evaluate effects of beta blocker on patients with TBI.

DETAILED DESCRIPTION:
The study will be conducted on polytrauma patient who are admitted from emergency room or postoperative with head trauma . Patients will be randomly assigned into two groups by sealed envelope technique into two equal groups.

Parameters assessment:

* Length of ICU stay
* Length of total hospital stay
* CT scan to exclude another intracranial hemorrhage or increase in hemorrhage
* Functional status will be assessed using the GCS
* Hemodynamic data ( bl.p / hr )
* Crystalloid volume that patient need in 24h
* Mortality rate

ELIGIBILITY:
Inclusion Criteria:

* GCS preoperative >10
* Abbreviated Injury Scale (AIS) >3
* Length stay in ICU >48 h

Exclusion Criteria:

* Hypersensitivity to propranolol
* Asthmatic patient
* COPD
* History of smoking
* Any cardiac problems eg: ( heart failure or HB )
* pheochromocytoma
* Pregnant patient
* Length stay <48h
* Death within 48 h of admission
* Patient who previously received any beta blocker at home.
* Symptomatic Bradycardia <60 b/m (sick sinus syndrome)
* Hemodynamic unstable patients

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
survival | 7 days
  number of surviving in patients receiving propranolol and patients who did not receive any beta blocker

SECONDARY OUTCOMES:
heart rate | 7 days
  number of patient showing effect of beta blocker on TBI related to HR
icu stay | 7 days
  number of patients were beta blocker in TBI affected on ICU and total hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: mostafa f mansour, MD, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Medicine, University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided